CLINICAL TRIAL: NCT02942589
Title: Effect of Portion-control Training on Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PortionSize103; R01DK059853 (NIH)
Record Dates: First submitted 2016-10-19; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Feeding Behaviors
Keywords: Portion Size
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 100% Portions (Experimental): Meal portion size: 100%
  Interventions: Other: Meal portion size
- 125% Portions (Experimental): Meal portion size: 125%
  Interventions: Other: Meal portion size
- 150% Portions (Experimental): Meal portion size: 150%
  Interventions: Other: Meal portion size
- 175% Portions (Experimental): Meal portion size: 175%
  Interventions: Other: Meal portion size

INTERVENTIONS:
Other: Meal portion size

SUMMARY:
The purpose of this study is to test whether food intake in response to large portion sizes differs between women who have received portion-control training and women who have not received such training. In a crossover design, women come to the laboratory on four occasions to eat a lunch of seven foods varying in energy density. Across meals, all foods are varied in portion size (100%, 125%, 150%, or 175% of baseline amounts). Food and energy intake is determined for each meal. Participants are from two groups: women who completed a one-year weight-loss trial in which they were trained in portion-control strategies, and women who had not received such training (community controls).

ELIGIBILITY:
Inclusion Criteria:

* Participant in the Portion-Control Strategies Trial (NCT01474759) OR
* Community control who regularly eats three meals per day

Exclusion Criteria:

* Score on the Eating Attitudes Test indicating symptoms of disordered eating
* Score on the Zung or Beck questionnaires indicating symptoms of depression
* Food allergies or restrictions
* Dislike for foods served in the study

Ages: 20 Years to 66 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Difference in energy intake across subject groups | Weeks 1, 2, 3, and 4
  Calculated energy intake (kcal) based on weight and energy density of food consumed
Difference in intake by weight across subject groups | Weeks 1, 2, 3, and 4
  Weights (grams) of all food consumed
Difference in energy density consumed across subject groups | Weeks 1, 2, 3, and 4
  Energy density (kcal/gram) of all food consumed

SECONDARY OUTCOMES:
Ratings of hunger and satiety across subject groups | Weeks 1, 2, 3, and 4
  100-point visual analog scales

OTHER OUTCOMES:
Ratings of food taste across subject groups | Week 5
  100-point visual analog scales
Ratings of food healthfulness across subject groups | Week 5
  100-point visual analog scales

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for the Study of Human Ingestive Behavior, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No